CLINICAL TRIAL: NCT04431531
Title: EMDR Pre-treatment Yoga for Complex Trauma Randomized Controlled Comparative Study
Brief Title: EMDR Pre-treatment Yoga for Complex Trauma
Acronym: YOGA-EMDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominique JANUEL (Other)
Responsible Party: Sponsor-Investigator, Dominique JANUEL, chief of Clinical Center Research, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10477M-YOGA-EMDR
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Trauma, Psychological
Keywords: Yogatherapy-EMDR-psychiatry
MeSH Terms: conditions — Psychological Trauma | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: the first group is about EMDR treatment. The second group is about YOGATHERAPY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yogatherapy-EMDR (Active Comparator): one of the two groups will have yogatherapy treatment and Eye movement desensibilization reprocessing (EMDR)
  Interventions: Other: 10 Sessions of yogatherapy associate with EMDR
- waiting list and EMDR (Active Comparator): The other group will have Eye movement desensibilization reprocessing
  Interventions: Other: The second group will have EMDR without yogatherapy

INTERVENTIONS:
Other: 10 Sessions of yogatherapy associate with EMDR — The first group will have Yogatherapy plus EMDR treatment
  Other Names: The second group will have EMDR without yogatherapy
  Arms: yogatherapy-EMDR
Other: The second group will have EMDR without yogatherapy — the second one will have EMDR treatment
  Arms: waiting list and EMDR

SUMMARY:
yoga is a technique of hope. Indeed, it is a practice that specifically combines postures, breathing technique and a state meditative. The combination of these elements produces multiple effects that are exposed to detailed in the publications of Bessel Van der Kolk (Price et al., 2017; Rhodes, Spinazzola, & van der Kolk, 2016; Van der Kolk, 2014; Van Der Kolk et al., 2014) and whose four main effects are summarized here:

* A regulation of the level of vigilance
* An improvement in self-awareness
* An increased sense of self-efficacy
* Improved metacognition, awareness and regulation emotional

DETAILED DESCRIPTION:
Yoga practice has shown benefits in treating multiple physical or mental disorders (Barnes, Bloom, & Nahin, 2008; Khalsa, 2004; Ross, Friedmann, Bevans, & Thomas, 2013) and has recently been evaluated for PTSD. We identified six randomized controlled studies measuring the effect of yoga in women (mostly) who experienced childhood violence (see table). With the exception of one pilot study (Dick, Niles, Street, Dimartino, & Mitchell, 2014; Mitchell et al., 2014), all studies show a significant reduction in PTSD symptoms compared to the pre-treatment period and compared to the control group (waiting list group). In particular, it was shown that this reduction in symptomatology was comparable to that of other commonly practiced psychotherapies, such as the exposure techniques of Behavioural and Cognitive Therapies or EMDR, and comparable to pharmacological treatments (Van Der Kolk et al., 2014). Prolonged yoga therapy would also significantly improve dissociative symptoms (Price et al., 2017). However, all these studies tested the effect of yoga therapy in isolation, without associating it with conventional and recommended treatments for trauma. However, given the fields of action of the yoga listed above, we think that it could be the ideal tool to prepare (in the pre-treatment phase) the work on traumatic memory. We believe that the combination of yoga therapy and EMDR would work in synergy to reduce complex PTSD and achieve a higher success rate than these individual approaches. In this work, we will use a yoga technique adapted to the treatment of psycho-trauma called "trauma sensitive yoga" (Emerson, 2015).

ELIGIBILITY:
Inclusion Criteria:

. Women

* Meets diagnostic criteria for Complex Post-traumatic Stress Disorder according to ICD-11 criteria, related to childhood sexual abuse
* PCL-5 must be at least 45
* Age between 18 and 70.
* Free, informed and signed consent.

Exclusion Criteria:

Neurological disorders

* Pregnant women
* Severe and/or unstable somatic diseases
* Diseases resulting in serious motor disorders (e.g. people paralyzed)
* Patient not affiliated with social security, State Medical Aid (AME)
* Patient hospitalized under stress in psychiatric care at the decision of the state representative or in psychiatric care at the request of a third party,
* Patient under guardianship, curatorship and protection of justice
* Patient participating in parallel biomedical research
* French language not mastered
* Persons unable to give consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female can participate to this study
Enrollment: 66 (Estimated)
Dates: Start 2016-09-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
PCL-5: Scale of post-traumatic stress disorder | first week
  PTSD Scale :
  Evaluation of clinical symptomatology and severity of PTSD
PCL-5: Scale of post-traumatic stress disorder | At twenty week
  PTSD Scale :
  Evaluation of clinical symptomatology and severity of PTSD

SECONDARY OUTCOMES:
CAPS-5: PTSD Scale Administered by Clinician | First week
  Evaluation of clinical symptomatology and severity of PTSD Diagnosis of comorbidities
CAPS-5: PTSD Scale Administered by Clinician | At ten week
  Evaluation of clinical symptomatology and severity of PTSD Diagnosis of comorbidities
CAPS-5: PTSD Scale Administered by Clinician | At twenty week
  Evaluation of clinical symptomatology and severity of PTSD Diagnosis of comorbidities

OTHER OUTCOMES:
CGI : Clinical global Impression | At first week
  Evaluation of overall clinical improvement.
CGI : Clinical global Impression | At ten week
  Evaluation of overall clinical improvement.
CGI : Clinical global Impression | At twenty week
  Evaluation of overall clinical improvement.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ch Ville Evrard, Neuilly-sur-Marne
  - Center for Psychotherapy and Psychotraumatology, Saint-Denis

IPD SHARING:
Plan to Share IPD: Undecided